CLINICAL TRIAL: NCT04461561
Title: Using Normalization Process Theory to Evaluate Providing Pediatric Palliative Care at End-of-Life as Web-Based Training Intervention for Nurses:
Brief Title: Using NPT to Evaluate Providing PPC as ELNEC-PPC WBT for Nurses
Acronym: ELNEC-PPC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Altoosi University College (Other)
Collaborators: Babylon University (Other)
Responsible Party: Principal Investigator, Moustafa Ali Ghazi Al-Shammari, Principal Investigator, Altoosi University College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AltoosiUC
Record Dates: First submitted 2020-06-28; First posted 2020-07-08 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Cancer; Cardiac Anomaly; Cystic Fibrosis; Muscular Dystrophy; HIV/AIDS; Batten's Disease; Cerebral Palsy
Keywords: life-limiting illnesses; pediatric palliative care; normalization process theory; End-of-life care; Web-Based Training Intervention
MeSH Terms: conditions — Neoplasms; Heart Defects, Congenital; Cystic Fibrosis; Muscular Dystrophies; Acquired Immunodeficiency Syndrome; Neuronal Ceroid-Lipofuscinoses; Cerebral Palsy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ELNEC-PPC WBT pluss usual care (Experimental): The End-of-Life Nursing Education Consortium (ELNEC) project is a national education initiative to improve nursing education on end-of-life care. The project is administered by the American Association of Colleges of Nursing and City of Hope National Medical Center. The intervention group received training through the Relais Academy website
  Interventions: Genetic: end-of-life nursing education consortium-pediatric palliative care as web based-training plus usual care
- Usual care only (No Intervention): Participants nurses deliver usual care as his/her role appropriate to neonates, infants, toddlers, preschoolers, school age, also to adolescents in selected unit of perinatal, neonatal, and settings which can be pediatric.

INTERVENTIONS:
Genetic: end-of-life nursing education consortium-pediatric palliative care as web based-training plus usual care — The End-of-Life Nursing Education Consortium (ELNEC) project is a national education initiative to improve nursing education on end-of-life care. The project is administered by the American Association of Colleges of Nursing and City of Hope National Medical Center. The intervention group received training through the Relais Academy website
  Other Names: ELNEC-PPC WBT course plus usual care
  Arms: ELNEC-PPC WBT pluss usual care

SUMMARY:
The purpose of this study is to explain the provision of palliative care at the end of life by the implementation of the ELNEC course, as WBT Program using the Normalization Process Theory, that focus attention on how complex interventions become routinely embedded in practice. In addition to, identify the changes implemented by the participant nurses (intervention group) in their clinical practice, after participating in WBT Program to provide Palliative Care alongside with usual care versus usual care only (control group) for children with life-limiting conditions or in the case of accidents/sudden death, at the end of life. And finally, provide findings that will assist in the interpretation of the trial results.

ELIGIBILITY:
Inclusion Criteria:

* The health care centers where the intervention will be administered include 1) Imam Sadiq (peace be upon him) Teaching Hospital; 2) Babylon Maternity and Children Teaching Hospital; 3) Al-Noor Hospital for Children; 4) Morgan Teaching Hospital, and 5) Babylon Oncology Center.
* The study population will be included all college nurses who completed their bachelor's degree and who have (master's or doctorate) degree in nursing sciences, that being employed for at least three months and not expected to be transferred to another unit within the study period during either morning or evening shifts and provides nursing care for both male and/or female of hospitalized patients 18 years.
* Use a computer (desktop or laptop) with access to the internet at home or work (phone line or internet access), or use a smartphone (with at least Android 6.0+ or iOS11. 0+) with internet access (Wi-Fi and/or mobile data) to join the online training course.
* Have a working email address and/or a working mobile number and have access to a computer or smartphone with internet access to complete questionnaires in a web browser.

Exclusion Criteria:

* Not interested.
* Not being employed for at least three months.
* Academic nurses who employed and continuing to work with other than selecting units, due to the carefully chosen only units that provide nursing care for both pediatric and adults or for pediatric, in order to achieve the study objectives.
* Enrolled in another experimental trial.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
The NoMAD Instrument, to describe respondents' experiences of using the intervention in the workplace. | 2 weeks after the end of WBT course
  The data collection instrument is NoMAD [1]. The NoMAD translated into Arabic for the purpose of evaluating the normalization of the pediatric palliative care provide by web-based training concept. The Arabic-NoMAD is divided into 3 sections. It begins with section A consisting of 12 questions about the respondent, section B with 3 general questions about the intervention. Section C contains 20 specific questions about the intervention, corresponding to the 4 constructs of the normalization process theory [2], with Coherence and Cognitive Participation has 4 items, 7 items for Collective Action, and 5 items for Reflexive Monitoring. The scale consists of 31 Likert-type items. Items in section B are answered with a 10-point Likert scale ranging from "Not at all" to "Completely". The items in part C are answered using a 5-point Likert scale, ranging from "Disagree Strongly" to 'Agree Strongly'. 'Neutral' and 'Not applicable'.
The NoMAD Instrument, to describe respondents' experiences of using the intervention in the workplace. | at 3 months for both groups
  The data collection instrument is NoMAD [1]. The NoMAD translated into Arabic for the purpose of evaluating the normalization of the pediatric palliative care provide by web-based training concept. The Arabic-NoMAD is divided into 3 sections. It begins with section A consisting of 12 questions about the respondent, section B with 3 general questions about the intervention. Section C contains 20 specific questions about the intervention, corresponding to the 4 constructs of the normalization process theory [2], with Coherence and Cognitive Participation has 4 items, 7 items for Collective Action, and 5 items for Reflexive Monitoring. The scale consists of 31 Likert-type items. Items in section B are answered with a 10-point Likert scale ranging from "Not at all" to "Completely". The items in part C are answered using a 5-point Likert scale, ranging from "Disagree Strongly" to 'Agree Strongly'. 'Neutral' and 'Not applicable'.

SECONDARY OUTCOMES:
The interview, using framework analysis, informed by normalization process theory toolkit | For 3-months post-course
  Semi-structured face-to-face interviews will be conducted by all nurses on how successful passing ELNEC-PPC WBT course from the selected setting. All participants had direct contact with patients. Three rounds of interviews will be conducted after 3 months. After consenting, participants will be interviewed by the main researcher (MA). All interviews will be audio-recorded and transcribed. They will be asked why they felt the change was significant. During the second round of interviews, will be asked about the most significant developments since the beginning of the program; they will be asked to share their views about pediatric palliative care and to describe the extent to which they were adopting the approach, and if not, why not. Topic guides were informed by NPT [3], it will be used the interactive NPT toolkit. It contains 16 questions, for thinking through an implementation problem. The work was embedding improved and edited statements and explanations into a web-enabled tool.

CONTACTS AND LOCATIONS:
Overall Officials: Nuhad Aldoori, Ph.D, Study Director — Babylon University/ Nursing Faculty; Amean A Yaser, Ph.D, Study Director — Babylon University/ Nursing Faculty
Locations (1):
- 1) Imam Sadiq (peace be upon him) Teaching Hospital; 2) Babylon Maternity and Children Teaching Hospital; 3) Al-Noor Hospital for Children; 4) Morgan Teaching Hospital; and 5) Babylon Oncology Center, Hillah, Babylon Province, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rapley T, Girling M, Mair FS, Murray E, Treweek S, McColl E, Steen IN, May CR, Finch TL. Improving the normalization of complex interventions: part 1 - development of the NoMAD instrument for assessing implementation work based on normalization process theory (NPT). BMC Med Res Methodol. 2018 Nov 15;18(1):133. doi: 10.1186/s12874-018-0590-y. PMID 30442093
- [Background] Rifkin LH, Stojadinovic S, Stewart CH, Song KH, Maxted MC, Bell MH, Kashefi NS, Speiser MP, Saint-Cyr M, Story MD, Rohrich RJ, Brown SA, Solberg TD. An athymic rat model of cutaneous radiation injury designed to study human tissue-based wound therapy. Radiat Oncol. 2012 May 8;7:68. doi: 10.1186/1748-717X-7-68. PMID 22568958
- [Background] May CR, Finch T, Ballini L, MacFarlane A, Mair F, Murray E, Treweek S, Rapley T. Evaluating complex interventions and health technologies using normalization process theory: development of a simplified approach and web-enabled toolkit. BMC Health Serv Res. 2011 Sep 30;11:245. doi: 10.1186/1472-6963-11-245. PMID 21961827
- [Derived] Al-Shammari MA, Yasir A, Aldoori N, Mohammad H. Using Normalization Process Theory to Evaluate an End-of-Life Pediatric Palliative Care Web-Based Training Program for Nurses: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2022 Nov 11;11(11):e23783. doi: 10.2196/23783. PMID 36367759
- See also: Related Info — http://www.normalizationprocess.org/npt-toolkit/